CLINICAL TRIAL: NCT02762149
Title: The Response Patterns to the Electrical Stimulation of Epidural Catheters With Varying Pulse Widths in Term Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analysis after 20 patients was convincing for a negative result for the primary outcome, so the study was stopped.
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-04
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Labor Pain
Keywords: Tsui Test; Labour; Epidural catheter
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.1ms pulse width (Active Comparator): The nerve stimulator will be connected to the epidural catheter through an adapter, which will be primed with a standard volume of 3 ml of sterile normal saline to allow for effective electrical conduction. The cathode terminal of the stimulator will then be attached to the metal hub of the adapter and the anode terminal will be connected to the electrode placed over the deltoid muscle. All patients will have the trans-catheter electric stimulation test (TCEST) performed with both a 1 ms pulse width and 0.1 ms pulse width and the order of administration will be randomized.
  Interventions: Device: Nerve stimulator
- 1ms pulse width (Active Comparator): The nerve stimulator will be connected to the epidural catheter through an adapter, which will be primed with a standard volume of 3 ml of sterile normal saline to allow for effective electrical conduction. The cathode terminal of the stimulator will then be attached to the metal hub of the adapter and the anode terminal will be connected to the electrode placed over the deltoid muscle. All patients will have the trans-catheter electric stimulation test (TCEST) performed with both a 1 ms pulse width and 0.1 ms pulse width and the order of administration will be randomized.
  Interventions: Device: Nerve stimulator

INTERVENTIONS:
Device: Nerve stimulator — The nerve stimulator (Stimpod NMS 450: Xavant technology (PTY) Ltd; Pretoria, South Africa or similar nerve stimulator) will be connected to the epidural catheter through an adapter (Johans ECG Adapter, Arrow International Inc., Reading). The epidural catheter and the adapter will be primed with a standard volume of 3 ml of sterile normal saline to allow for effective electrical conduction. Secured connections and avoidance of any air within in the system must be ensured to avoid high impedance in the circuit, which could result in false negatives. The cathode terminal of the stimulator will then be attached to the metal hub of the adapter and the anode terminal will be connected to the electrode placed over the deltoid muscle.
  Other Names: Stimpod NMS 450

SUMMARY:
Epidural analgesia is commonly used for labor pain relief due to its safety and effectiveness. Despite a very high success rate, the epidural technique remains a somewhat blind technique and failures continue to occur. Unfortunately, there are no imaging techniques that can be used at the bedside to determine the proper positioning of the epidural catheter. The trans-catheter electric stimulation test (TCEST) has been successfully used for this purpose. This test is occasionally performed in situations where the immediate confirmation of the proper epidural catheter location is deemed necessary. The test helps to predict which epidurals might fail so that appropriate measures could be immediately implemented.

There has been one duration of electrical stimulus (0.2 milliseconds) that has been used in the majority of studies and in clinical practice. With this duration of stimulation, the vast majority of cases show a unilateral motor response of the lower limbs during the TCEST. Studies on the stimulation of peripheral nerves (nerves in the arms and legs) have shown that an electrical stimulus with a longer duration is able to stimulate nerves which are farther away. Since nerves in the epidural space are similar in composition to peripheral nerves, the investigators expect to see a higher rate of bilateral response with the longer duration of stimulus. The investigators also hope to show that this bilateral response is predictive of a better functioning epidural.

The investigators hypothesize that the incidence of a bilateral response to the TCEST will be higher with the 1.0 ms pulse width compared to 0.1 ms pulse width. Furthermore, the investigators hypothesize that a bilateral motor response associated with the 1.0 ms pulse width will be predictive of symmetry of sensory and motor block and of lower consumption of local anesthetic.

DETAILED DESCRIPTION:
This will be a randomized double-blind controlled study. After recruitment of the patient, epidural anesthesia will be performed in the standard fashion employed in the investigators' institution by a fellow or staff. Spinal ultrasound will be used prior to performing the epidural catheter insertion. The trans-catheter electric stimulation test (TCEST) will be performed at both a 0.1ms pulse width and a 1ms pulse width. The order in which the two pulse widths are applied will be randomly decided by computer. The test dose of local anesthetic will then be administered, and the TCEST will be repeated 5 minutes later. Again, both pulse widths (0.1ms, 1ms) will be used, and the order in which they are applied will be decided randomly.

Following the second testing, a loading dose of the standard anesthetic solution will be administered. The sensory level to ice will be tested at 20 minutes following injection of the loading dose of bupivacaine and fentanyl. The sensory level will be assessed from the sacral to the thoracic levels, bilaterally. The motor response pattern will be recorded for all TCESTs performed, and any relationship between pulse width and response pattern will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Women 16 years of age and older requesting an epidural for labour analgesia
* Ability to communicate in English
* Informed consent

Exclusion criteria:

* Refusal to provide written informed consent
* Inability to communicate in English
* Abnormal vertebral anatomy, including but not limited to previous spine surgery and scoliosis
* Allergy or hypersensitivity to lidocaine, bupivacaine or fentanyl
* Coexisting neurological disorders
* Implanted electronic devices

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Motor response pattern | 5 minutes
  Motor response pattern to the electrical stimulation of the epidural catheter, either unilateral or bilateral.

SECONDARY OUTCOMES:
Sensory level | 2 hours
  The sensory level to ice at 20 minutes and 2 hours following injection of the standard epidural loading dose. The sensory level will be assessed from the sacral to the thoracic levels, bilaterally.
Motor block | 2 hours
  Lower extremity motor block as assessed by the Bromage score (Range: 0-3) bilaterally at 20 minutes and 2 hours following the loading dose.
  0 = No motor block (full flexion of knees and feet)
  1. = Partial motor block (just able to move knees and feet)
  2. = Almost complete motor block (able to move feet only)
  3. = Complete motor block (unable to move feet or knees)
Current (mA) | 5 minutes
  The current required to elicit a motor response on the initial TCEST and at 5 minutes after the test dose
Consumption of local anesthetic | 2 hours
  Amount of local anesthetic consumed as measured on the pump in the first 2 hours.
Epidural block failure | 2 hours
  Failure of the epidural analgesia, defined as no evidence of a sensory block to ice and absent pain relief in the first 20 minutes, OR the need for epidural catheter replacement within 2 hours of the loading dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zakus P, Bittencourt R, Downey K, Tsui BCH, Carvalho JCA. The effect of an increased pulse width on the pattern of motor response (unilateral versus bilateral) during the Tsui test in labouring parturients: a randomized crossover trial. Can J Anaesth. 2017 Dec;64(12):1211-1217. doi: 10.1007/s12630-017-0977-y. Epub 2017 Sep 21. PMID 28936608